CLINICAL TRIAL: NCT06622434
Title: New Adjuvant Vaccine in Glioblastoma, a Phase 1/2a Study (NAVIG-1)
Brief Title: New Adjuvant Vaccine in Glioblastoma, a Phase 1/2a Study
Acronym: NAVIG-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP240512; 2024-514567-26-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-25; First posted 2024-10-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Newly Diagnosed Glioblastoma
Keywords: Cancer vaccine; Glioblastoma; Telomerase; TERT; PTPRZ1; Immunomodulation
MeSH Terms: conditions — Glioblastoma | interventions — Immunization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A52-Mel/A49-Mel/Li28 (Experimental): One month after completion of concurrent radiochemotherapy, patients will be immunized during the adjuvant phase of monthly temozolomide with subcutaneous injections of the vaccine formulation (D0, W2, W4, W6, and then every 2 months until progression) consisting of 2 tumor antigens (TERT and PTPRZ1) adjuvanted with synthetic melanin and a TLR9 agonist (CpG-ODN).
  Interventions: Biological: immunization

INTERVENTIONS:
Biological: immunization — One month after completion of concurrent radiochemotherapy, patients will be immunized during the adjuvant phase of monthly temozolomide with subcutaneous injections of the vaccine formulation (D0, W2, W4, W6, and then every 2 months until progression) consisting of 2 tumor antigens (TERT and PTPRZ1) adjuvanted with synthetic melanin and a TLR9 agonist (CpG-ODN).

SUMMARY:
This phase I/II trial evaluates the safety and the immunological efficacy of a cancer vaccine against 2 glioma-associated antigens in newly-diagnosed glioblastomas. All patients enrolled in the study will receive standard treatment consisting of surgical resection of the tumor followed by radio-chemotherapy. Immunotherapy will begin 4 weeks after the completion of radiotherapy.

DETAILED DESCRIPTION:
This therapeutic vaccine targeting 2 identified glioma-associated antigens (TERT and PTPRZ1) is based on a new formulation that contains synthetic melanin and a TLR9 agonist, which is caable to induce strong cellular immune responses.

One month after glioblastoma patients have completed the initial phase of treatment with concurrent radiochemotherapy, patients will be immunized during the adjuvant phase of monthly temozolomide. Immunizations will follow the standard schedule of a priming phase (D0, W2, W4, and W6) followed by a boost phase with one immunization every 2 months for a total of 12 months.

Phase 1: subcutaneous injections at one of 3 pre-specified dose levels of peptides Phase 2a: subcutaneous injections at the dose selected in the phase 1 part. Safety will be evaluated clinically and with blood samples at each treatment visit. Efficacy will be assessed with anti-PTPRZ1 and anti-TERT specific T cell responses in peripheral blood, and with cerebral MRI every other months

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years old
* free, informed and written consent signed
* Histologically confirmed glioblastoma
* Patients previously treated with concurrent radiotherapy (at least 45 Gy) with concomitant temozolomide, before the beginning of the 6 additional monthly cycles of temozolomide. Radiation therapy must have been completed 28 to 45 days prior to the first study treatment
* Karnofsky Performance Status ≥ 60%
* Patients must be human leukocyte antigen (HLA)-A2 positive.
* PTPRZ1 expression in the tumor
* Available tumor tissue for post hoc (retrospective) assessment of TERT promoter mutations and MGMT promoter methylation status
* Life expectancy ≥ 3 months
* Adequate organ function laboratory values within 15 days before initiation of treatment (see table in section 6.1)
* Women or Male of childbearing potential (WOCBP) must use contraceptive methods during and for 180 days after the last dose of temozolomide or up to 120 days after the last dose of vaccine, whichever is longer (see section 6.3). No sperm donation during the study and until 7 months after the end of the treatment period.
* Patient affiliated to the social security scheme

Exclusion Criteria:

* Known extracranial metastatic or leptomeningeal disease
* Grade 4 astrocytoma IDH mutant
* Steroid requirement >10 mg prednisone daily (or equivalent) at time of inclusion
* Patients with prior malignancy active within the last 3 years
* Patients receiving immunomodulatory or immunosuppressive therapy
* Carmustine wafers (GliadelR) implantation during surgery
* Phase 1 only: patient eligible and willing to be treated with Optune (TTF fields)
* History of autoimmune disease (lupus, rheumatoid arthritis, inflammatory bowel disease...)
* Previous treatment with bevacizumab or other Vascular Endothelial Growth Factor (VEGF) antagonists
* Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection within the previous 4 weeks or requirement for intravenous (IV) antibiotics within the last two weeks
* Breast-feeding or pregnant women.
* Contra-indications to IRM
* Contra-indications to investigational medicinal product and/or to auxiliary medicinal products
* Participation to another interventional clinical trial, clinical investigation or another interventional study or being in the exclusion period at the end of a previous study
* Patient unable to follow the procedures and constraints of the protocol
* Patient under legal protection (protection of the court, or in curatorship or guardianship).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-05-08 (Estimated); Study Completion 2027-05-08 (Estimated)

PRIMARY OUTCOMES:
safety/efficacy | 12 months
  - phase 1: to assess the maximum tolerated dose (MTD)
safety/efficacy | 2 months
  - phase 2a : to assess anti-PTPRZ1/ TERT specific T cell responses

SECONDARY OUTCOMES:
Overall survival | 12 months
  The time interval from the start of treatment to the date of death from any cause.
Progression free survival | 12 months
  Tumor response will be assessed using RANO 2.0 criteria
the evaluation of quality of life | 5 months
  EORTC-QLQC30 questionnaire and BN20 module will be completed by each patient (Not all= 1; A little=2; Quite a bit= 3 ; Very Much=4)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CARPENTIER, Pr, Study Chair — APHP- Hôpital Saint Louis
Locations (1):
- Department of Neurology, Hopital Saint louis (APHP), Paris, France